CLINICAL TRIAL: NCT04775069
Title: A Prospective Study Comparing the Antibody Response of Subjects With Chronic Liver Disease to mRNA, Inactivated Virus and Adenovirus Vector COVID-19 Vaccines
Brief Title: Antibody Response to COVID-19 Vaccines in Liver Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHCTC_COVID-19_VACCINE_Ab
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — BNT162 Vaccine; sinovac COVID-19 vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mRNA Group (Active Comparator): The subjects will be vaccinated with the mRNA vaccine (Pfizer-Biontech).
  Interventions: Biological: BNT162b2
- Inactivated Virus Group (Active Comparator): The subjects will be vaccinated with inactivated SARS Cov-2 (Sinovac).
  Interventions: Biological: CoronaVac
- Adenovirus-vector Group (Active Comparator): The subjects will be vaccinated with adenovirus-vector COVID-19 vaccine (Astrazeneca-Oxford).
  Interventions: Biological: AZD1222

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular injection
  Arms: mRNA Group
Biological: CoronaVac — Intramuscular injection
  Arms: Inactivated Virus Group
Biological: AZD1222 — Intramuscular injection
  Arms: Adenovirus-vector Group

SUMMARY:
Currently the Pfizer-Biontech (mRNA), Sinovac (inactivated virus) and Astrazeneca-Oxford (adenovirus-vector) COVID-19 vaccines are available for vaccination in HK. The American Association of Liver Disease has recently published consensus statements for COVID-19 vaccination in subjects with chronic liver disease (CLD). Patients with CLD have dysregulated innate and adaptive immune response that may be associated with vaccine hypo-responsiveness and there are no data as to whether these patients may respond differently to the various vaccines. The Humanity and Health Medical Center (HHMC) is an active participant of the HK government COVID-19 vaccination programs and patients with CLD follow-up at HHMC will have access to the three different vaccines. The aim of this prospective study is to compare the antibody response of CLD subjects to the Pfizer-Biontech (mRNA), Sinovac (inactivated virus) and Astrazeneca-Oxford (adenovirus-vector) COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with chronic liver disease (CLD) at the Humanity and Health Medical Group and eligible for the HK government vaccination programme;
2. Able to understand and sign informed consent.;
3. Underlying CLD- defined as patients with chronic hepatitis B or C infections, liver cirrhosis, metabolic associated liver disease, hepatocellular carcinoma, alcoholic liver disease, autoimmune hepatitis, hemochrombtosis.

Exclusion Criteria:

1. Patients contraindicated for the COVID -19 Vaccination Program due to uncontrolled co-morbitities;
2. Past allergies to other vaccines;
3. Pregnant subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Antibody response | at 4 weeks after second dose
  Covid-19 Antibodies IgG titres at 4 weeks after second dose

SECONDARY OUTCOMES:
Antibody response | at one year after second dose
  Covid-19 Antibodies IgG titres at one year after second dose

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity & Health Medical Group Limited, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fix OK, Blumberg EA, Chang KM, Chu J, Chung RT, Goacher EK, Hameed B, Kaul DR, Kulik LM, Kwok RM, McGuire BM, Mulligan DC, Price JC, Reau NS, Reddy KR, Reynolds A, Rosen HR, Russo MW, Schilsky ML, Verna EC, Ward JW, Fontana RJ; AASLD COVID-19 Vaccine Working Group. American Association for the Study of Liver Diseases Expert Panel Consensus Statement: Vaccines to Prevent Coronavirus Disease 2019 Infection in Patients With Liver Disease. Hepatology. 2021 Aug;74(2):1049-1064. doi: 10.1002/hep.31751. PMID 33577086
- [Background] Mulligan MJ, Lyke KE, Kitchin N, Absalon J, Gurtman A, Lockhart S, Neuzil K, Raabe V, Bailey R, Swanson KA, Li P, Koury K, Kalina W, Cooper D, Fontes-Garfias C, Shi PY, Tureci O, Tompkins KR, Walsh EE, Frenck R, Falsey AR, Dormitzer PR, Gruber WC, Sahin U, Jansen KU. Phase I/II study of COVID-19 RNA vaccine BNT162b1 in adults. Nature. 2020 Oct;586(7830):589-593. doi: 10.1038/s41586-020-2639-4. Epub 2020 Aug 12. PMID 32785213
- [Background] Zhang Y, Zeng G, Pan H, Li C, Hu Y, Chu K, Han W, Chen Z, Tang R, Yin W, Chen X, Hu Y, Liu X, Jiang C, Li J, Yang M, Song Y, Wang X, Gao Q, Zhu F. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine in healthy adults aged 18-59 years: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Feb;21(2):181-192. doi: 10.1016/S1473-3099(20)30843-4. Epub 2020 Nov 17. PMID 33217362
- [Background] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298